CLINICAL TRIAL: NCT02466958
Title: Double-blind Placebo-controlled Trial of Levomilnacipran in Geriatric Depression
Brief Title: Trial of Levomilnacipran in Geriatric Depression
Acronym: LMIL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Helen Lavretsky, MD, Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IIT-USA-000620
Record Dates: First submitted 2015-05-29; First posted 2015-06-09 (Estimated); Results first posted 2019-04-26 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Major Depressive Disorder
Keywords: depressed; older adults; antidepressants; depression; MDD
MeSH Terms: conditions — Depressive Disorder, Major; Consciousness Disorders; Depression | interventions — Levomilnacipran

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- levomilnacipran (FETZIMA) (Active Comparator): All eligible subjects will be randomized to levomilnacipran or placebo group using a computer-generated random assignment scheme, which assigned subjects in a 1:1 ratio to each group. Randomization will be done prior to subject's being assigned to the groups.
  Interventions: Drug: levomilnacipran
- Placebo (Placebo Comparator): All eligible subjects will be randomized to levomilnacipran or placebo group using a computer-generated random assignment scheme, which assigned subjects in a 1:1 ratio to each group. Randomization will be done prior to subject's being assigned to the groups.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: levomilnacipran — antidepressant
  Other Names: FETZIMA
  Arms: levomilnacipran (FETZIMA)
Drug: Placebo — an inactive drug
  Other Names: inactive substance
  Arms: Placebo

SUMMARY:
The purpose of this study is to examine the effects of levomilnacipran (FETZIMA) compared to placebo for the treatment of depression in older adults.

DETAILED DESCRIPTION:
A 12-week pilot double-blind comparison of levomilnacipran (FETZIMA) to placebo for the treatment of geriatric depression. The investigators are interested in assessing the efficacy of levomilnacipran (LMIL) to placebo (PBO), and exploring the effects of antidepressant response on brain connectivity and neuroplasticity. This pilot study is designed to determine any differences in the efficacy, safety and tolerability of levomilnacipran compared to placebo, and to perform dose finding (20-120 mg per day) in 40 older depressed adults. The investigators anticipate that the LMIL will be superior to PBO in improving levels of depressive symptoms and rates of remission, as well as improving cognition, apathy, and quality of life. This proposal expands the investigator's focus on the biomarkers of neuroplasticity that have been used in several prior studies and demonstrated responsivity to antidepressant treatment. The purpose is to examine this directly in 40 older adults with major depression. This proposed trial will also serve as a pilot study to estimate the efficacy and tolerability of the drug in older depressed adults, and the dose-finding in this population.

ELIGIBILITY:
Inclusion Criteria:

* 60 years of age or older
* The presence of a major depressive disorder diagnosed according to the Diagnostic and Statistical Manual and Mental Disorders, 5th edition (DSM-V) criteria
* A 24-item Hamilton Rating Scale for Depression (HAMD) score of 16 or higher at baseline
* Mini-Mental State Exam (MMSE) score > 24.

Exclusion Criteria:

Subjects will be excluded if they had 1) any current and/or lifetime history of other psychiatric disorders (except unipolar depression with or without comorbid generalized anxiety disorder), or 2) recent unstable medical or neurological disorders; 3) any disabilities preventing participation in the study or in the MRI; 4) diagnosis of dementia; 5) acute suicidality; 6) subjects with known allergic reactions to milnacipran, uncontrolled narrow angle glaucoma, seizures, poorly-controlled hypertension or ischemic changes on ECG, serotonin syndrome, or the recently used monoamine oxidase inhibitors (MAOIs) within last 4 weeks; 7) ineligible for MRI (e.g., metal in the body or claustrophobia)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2016-06; Primary Completion 2018-12-09 (Actual); Study Completion 2018-12-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Helen Lavretsky, M.D., Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Semel Institute - Neuropsychiatric Institute (NPI), Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Krause-Sorio B, Kilpatrick L, Siddarth P, Ercoli L, Laird KT, Aguilar-Faustino Y, Milillo MM, Narr KL, Lavretsky H. Cortical thickness increases with levomilnacipran treatment in a pilot randomised double-blind placebo-controlled trial in late-life depression. Psychogeriatrics. 2020 Mar;20(2):140-148. doi: 10.1111/psyg.12475. Epub 2019 Jul 22. PMID 31332902
- [Derived] Lee SM, Dong TS, Krause-Sorio B, Siddarth P, Milillo MM, Lagishetty V, Datta T, Aguilar-Faustino Y, Jacobs JP, Lavretsky H. The intestinal microbiota as a predictor for antidepressant treatment outcome in geriatric depression: a prospective pilot study. Int Psychogeriatr. 2022 Jan;34(1):33-45. doi: 10.1017/S1041610221000120. Epub 2021 Mar 24. PMID 33757609

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Levomilnacipran (FETZIMA) | Placebo
Started | 17 | 12
Completed | 7 | 9
Not Completed | 10 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Levomilnacipran (FETZIMA) | Placebo | Total
Number analyzed (Participants) | 17 | 12 | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 4 | 4
  >=65 years | 17 | 8 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.24 (4.6) | 69.08 (6.6) | 71.5 (5.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 8 | 18
  Male | 7 | 4 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 16 | 8 | 24
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 17 | 12 | 29
Hamilton Depression Rating Scale Score [Mean (Standard Deviation); unit: units on a scale] — This measure includes 24 items. Response options vary item to item and include the following ranges: [0-2], [0-3], and [0-4]. A score of 0 suggests absence of symptoms and/or difficulties and higher scores represent more severe difficulties. Possible overall score range [0-74], higher scores representing more severe difficulties.
  units on a scale | 17.88 (2.5) | 19.92 (2.6) | 18.7 (2.7)

OUTCOME MEASURES:

1. Primary Outcome: Hamilton Depression Rating Scale (HDRS) Scores 24
Description: This measure includes 24 items. Response options vary item to item and include the following ranges: [0-2], [0-3], and [0-4]. A score of 0 suggests absence of symptoms and/or difficulties and higher scores represent more severe difficulties. Possible overall score range [0-74], higher scores representing more severe difficulties.
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Levomilnacipran (FETZIMA) | Placebo
Number analyzed (Participants) | 17 | 12
units on a scale
  Baseline | 17.88 (2.5) | 19.92 (2.6)
  12 Weeks | 6.86 (5.7) | 10.33 (7.1)

2. Secondary Outcome: Clinical Global Impression Scale (CGI) Scores
Description: 7-Point Likert Scale [1 = very much improved, 2 = much improved, 3 = minimally improved, 4 = no change, 5 = minimally worse, 6 = much worse, 7 = very much worse].
Time Frame: Week 12 reported
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Levomilnacipran (FETZIMA) | Placebo
Number analyzed (Participants) | 7 | 9
units on a scale | 3.00 (.81) | 3.33 (1.11)

3. Secondary Outcome: Geriatric Depression (GDS) Scores
Description: The GDS has a total of 30 items with response options [Yes/No]. Total score range is [0-30]. Higher scores represent more severe difficulties.
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Levomilnacipran (FETZIMA) | Placebo
Number analyzed (Participants) | 17 | 12
units on a scale
  Baseline | 13.5 (4.0) | 15.33 (4.8)
  12 Weeks | 11.71 (5.6) | 11.33 (3.6)

ADVERSE EVENTS:
Time Frame: 09/2016 - 07/2018; 1 years and 10 months
Arm/Group | Levomilnacipran (FETZIMA) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/12
Other Adverse Events (participants affected / at risk) | 11/17 | 2/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Levomilnacipran (FETZIMA) (N=17) | Placebo (N=12)
Teeth grinding (Musculoskeletal and connective tissue disorders) | 3 | 0
Sleepiness (Psychiatric disorders) | 1 | 0
Decreased duration of sleep (Psychiatric disorders) | 2 | 0
Reduced salivation (General disorders) | 2 | 1
Sweating (General disorders) | 1 | 0
Falls (Musculoskeletal and connective tissue disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 4 | 0
Upset stomach (Gastrointestinal disorders) | 1 | 0
Micturition disturbance (Renal and urinary disorders) | 6 | 0
Orthostatic dizziness (General disorders) | 1 | 1
Orgastic dysfunction (Reproductive system and breast disorders) | 1 | 0
Increased blood pressure (Cardiac disorders) | 1 | 1
Heart palpitations/tachycardia (Cardiac disorders) | 3 | 0
Visual disturbances (General disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-11-30): https://cdn.clinicaltrials.gov/large-docs/58/NCT02466958/Prot_SAP_000.pdf